CLINICAL TRIAL: NCT04794660
Title: The Study for the "Cervical Cancer Screening and Treatment Algorithms Study Using HPV Testing in Africa"
Acronym: CESTA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: International Agency for Research on Cancer (Other)
Collaborators: World Health Organization (Other); University of KwaZulu (Other); Cheikh Anta Diop University, Senegal (Other); Walter Sisulu University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: CESTA / PP202104-08
Record Dates: First submitted 2021-02-16; First posted 2021-03-12 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: HPV Infection
Keywords: VIA triage; HIV serostatus
MeSH Terms: conditions — Papillomavirus Infections | interventions — Human Papillomavirus DNA Tests; Colposcopy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Masking Description: Care providers and participants are masked to the intervention ahead of the intervention. However, the strategy delivery is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1 (Active Comparator): In this arm, HPV-positive women will undergo a Visual Inspection with Acetic Acid (VIA) triage test followed by biopsies. Treatment by thermal ablation (or cryotherapy in South Africa) will be applied to VIA positive women eligible for ablative treatment. Non eligible women will be referred to colposcopy.
  Interventions: Diagnostic Test: HPV DNA Test; Diagnostic Test: VIA triage test; Procedure: Treatment by ablative treatment; Procedure: Colposcopy
- Arm 2 (Active Comparator): In this arm, HPV positive women will get biopsies and receive an ablative treatment by thermal ablation (or cryotherapy in South Africa) if they are eligible to ablative treatment. Non eligible women will be referred to colposcopy
  Interventions: Diagnostic Test: HPV DNA Test; Procedure: Treatment by ablative treatment; Procedure: Colposcopy

INTERVENTIONS:
Diagnostic Test: HPV DNA Test — Screening for HPV using a HPV DNA test
Diagnostic Test: VIA triage test — VIA is a technique in which cervical neoplastic lesions are visually diagnosed after application of 3-5% acetic acid without using any magnification device.
  After application of 3 - 5% acetic acid, using the naked eye, the cervix is examined for the presence of an aceto-white lesion located in the transformation zone. The results are classified as either positive or negative, inadequate or suspicion of cancer
  Arms: Arm 1
Procedure: Treatment by ablative treatment — Cryotherapy or Thermal Ablation are performed on the cervix.
Procedure: Colposcopy — Colposcopy visit are offered to women with non visible squamous columnar junction or ineligible for ablative treatment.

SUMMARY:
The main objectives of CESTA are (1) to compare the efficacy of two cervical cancer screening algorithms: HPV test followed by visual inspection with acetic acid (VIA) and treatment (HPV + VIA + treat) and HPV test followed by immediate treatment (HPV + treat). The study will be conducted to address its objectives in women living with HIV (from now on called HIV positive women); and 2) To evaluate the performance of other techniques for primary screening and as triage for HPV positives WLHIV.

1,500 women living with HIV WLHIV will be recruited from HIV care clinics, also called antiretrovirals (ARV) clinics in South Africa. After giving informed consent, women will be screened with HPV testing and those that have a HPV positive test will be randomized at a 4:1 ratio into HPV + VIA + treat (Arm 1) and HPV + treat (Arm 2). Women in Arm 1 will receive VIA and only positive for VIA will be treated. In Arm 2, all HPV positive women will be treated. Women that are eligible for ablative treatment will be randomized into treatment with TA or cryotherapy in both arms. Others will be referred to colposcopy. After VIA in Arm 1 or before treatment in Arm 2, the nurses will collect 2-4 biopsies on all HPV positive women. The biopsies will be used as gold standard for disease detection. Treated women will be called by telephone after 1 week and 1 month to assess side-effects and satisfaction with the procedures. Cervical samples from women will be tested with HPV DNA test and HPV mRNA test to evaluate different screening tests for WLHIV. All women with a positive HPV test (treated or not) will be called back after 1 year for a follow-up visit. At this visit, women will be screened with HPV testing and VIA and 2-4 colposcopy-directed biopsies will be taken from all HPV positive women. Women with remaining/recurrent CIN2+ disease will receive appropriate management.

ELIGIBILITY:
Inclusion Criteria:

* Willing to disclose HIV status
* HIV negative women aged 30-54 years; HIV positive women aged 25-54 years
* Mentally competent to give informed consent
* Physically able to have a pelvic exam

Exclusion Criteria:

* Women reporting no previous sexual activity
* History of cervical cancer
* Treatment for cervical precancer in the last six months
* Hysterectomy
* Pregnancy
* Serious pre-existing medical conditions (e.g. history of bleeding disorders, serious physical or mental disease)

Ages: 25 Years to 54 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1500 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of women treated with high grade lesions in both arms | up top 1 month
Percentage of women treated with low grade lesions in both arms | up to 1 month

SECONDARY OUTCOMES:
Persistence of HPV infection and lesions at one year | up to 14 months
  all HPV positive women at screening will be asked to come back at one year to be tested for HPV. HPV positive women at one year will be refered to colposcopy and biopsies will be taken

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie Broutet, Dr, Principal Investigator — World Health Organization; Maribel Almonte, Dr, Principal Investigator — IARC
Locations (3):
- Roi Baudoin hospital, Dakar, Senegal
- South Africa (2):
  - Wentworth Hospital, Durban
  - Frere Hospital, East London

DOCUMENTS (2):
  • Study Protocol (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT04794660/Prot_000.pdf
  • Informed Consent Form (2019-06-11): https://cdn.clinicaltrials.gov/large-docs/60/NCT04794660/ICF_001.pdf